CLINICAL TRIAL: NCT06048978
Title: The Effect of Starch Processing on Postprandial Blood Glucose in Humans
Brief Title: Blood Glucose Response of Processed Starch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INQUIS Clinical Research (Industry)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: INQ-2330
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Glycemic Response
Keywords: Postprandial Glycemia; Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Native Starch, then Processed Starch (Experimental): Participants will first receive the Commercial Native Starch in a fasting state in one clinical visit. After a washout of >24 hours, the participants will then receive the Extrusion Processed Starch in a fasting state in one clinical visit.
  Interventions: Other: Commercial native starch without processing; Other: Modified starch with extrusion processing
- Processed Starch, then Native Starch (Experimental): Participants will first receive the Extrusion Processed Starch in a fasting state in one clinical visit. After a washout of >24 hours, the participants then will receive the Commercial Native Starch in a fasting state in one clinical visit.
  Interventions: Other: Commercial native starch without processing; Other: Modified starch with extrusion processing

INTERVENTIONS:
Other: Commercial native starch without processing — A food-grade commercial native starch without processing that has been rehydrated into a pudding for oral consumption.
Other: Modified starch with extrusion processing — A food-grade modified starch with extrusion processing that has been rehydrated into a pudding for oral consumption.

SUMMARY:
The goal of this clinical trial is to determine the postprandial glycemic response of the two starches in humans. Participants will be asked to consume 2 test foods on 2 separate occasions and provide blood glucose samples over 120 minutes postprandial.

DETAILED DESCRIPTION:
Enrolled participants who are generally healthy and free of major chronic conditions will be randomized to receive either Commercial Native Starch or Extrusion Processed Starch first and then will be crossed over to receive the opposite Intervention. The study will consist of two clinical test visits of 120 minutes separated by a washout period of at least 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* adult males or non-pregnant females.
* eligible to receive income in Canada.

Exclusion Criteria:

* age less than 18 years
* any known food allergies or intolerances to the investigational product
* medications known to affect glucose tolerance -but stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable
* known history of diabetes mellitus or the use of anti-hyperglycemic drugs or insulin to treat diabetes and related conditions
* any major medical or surgical events requiring hospitalization within the preceding 3 months
* the presence of disease or drug(s) which influence digestion and absorption of nutrients
* the short-term use of systemic steroids or atypical antipsychotics (<4 weeks) (all of which have major effects on glucose and metabolism and body fat distribution)
* any other medications or conditions which might, in the opinion of the Medical Director of INQUIS Clinical Research Ltd. (INQUIS), either 1) make participation dangerous to the subject or to others, or 2) affect the results
* any subject who cannot or will not comply with the experimental procedures or do not follow INQUIS safety guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Postprandial Glycemia | -5 to 120 minutes after intervention administration
  Incremental area under the curve for blood glucose over 120 minutes.

SECONDARY OUTCOMES:
Incremental Blood Glucose | 0, 15, 30, 45, 60, 90, and 120 minutes after intervention administration
  Change in blood glucose from baseline at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, DM (Oxon), Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No